CLINICAL TRIAL: NCT01513785
Title: New Dual Therapy for Primary Treatment of Helicobacter Pylori Infection：a Pilot Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiaobo Li, Xiaobo Li, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rjyyxhk0904
Record Dates: First submitted 2012-01-16; First posted 2012-01-20 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Functional Dyspepsia
Keywords: H. pylori; Dual therapy; Amoxicillin; Rabeprazole
MeSH Terms: interventions — Rabeprazole; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- group R20A (Active Comparator): All the patients were sent to a penicillin skin test before treatment except they were given penicillin before. The group R20A will receive 14 days of Amoxicillin 1g t.i.d and Rabeprazole 20 mg b.i.d. PPI was taken 30 minutes before meals while antibiotic was taken 30 minutes after meals.
  Interventions: Drug: Amoxicillin and Rabeprazole
- group R10A (Active Comparator): All the patients were sent to a penicillin skin test before treatment except they were given penicillin before. The group R10A will receive 14 days of Amoxicillin 1g t.i.d and Rabeprazole 10 mg b.i.d. PPI was taken 30 minutes before meals while antibiotic was taken 30 minutes after meals.
  Interventions: Drug: Rabeprazole and Amoxicillin

INTERVENTIONS:
Drug: Rabeprazole and Amoxicillin — Amoxicillin (Zhuhai United Laboratories Co., Zhuhai, China) 1g t.i.d and Rabeprazole (Misato Plant of Eisai Co., Ltd. Japan) 10 mg b.i.d.for 14 days.
  Other Names: Amoxycillin Capsules; Sodium Rabeprazole Enteric-coated Tablets
  Arms: group R10A
Drug: Amoxicillin and Rabeprazole — Amoxicillin (Zhuhai United Laboratories Co., Zhuhai, China) 1 g t.i.d and Rabeprazole (Misato Plant of Eisai Co., Ltd. Japan) 20 mg b.i.d. for 14 days
  Other Names: Amoxycillin Capsules; Sodium Rabeprazole Enteric-coated Tablets
  Arms: group R20A

SUMMARY:
The efficacy of traditional triple therapy has been decreased to such an unacceptable level as 70% in many areas. The study is based on the hypothesis: the most important factors which influence the effect of Helicobacter pylori (H. pylori) eradication included acid suppression intensity and sensitivity of antibiotics. So the investigators chose dual therapy because it is simple and verified to be useful. Rabeprazole, as a new proton pump inhibitor (PPI), is reported to be less susceptible to the influence of genetic polymorphisms for CYP2C19. So it has a greater and faster acid suppression effect compared to other PPIs. Amoxicillin is one of effective antibiotics to H. pylori with few side effects. The antibiotic resistance of Amoxicillin is no more than 3% in China. The purpose of our trial is to evaluate and compare the efficacy and safety of dual therapy regimens with different doses of Rabeprazole for initial treatment of H. pylori infection.

DETAILED DESCRIPTION:
The current recommended triple regimen for H. pylori treatment provides unacceptable low success rates because of high antibiotic resistance and poor compliance. Dual therapy had been used before and can be modified to get good eradication rate. The aim of our trial is to evaluate and compare the efficacy and safety of dual therapy regimens for initial treatment of H. pylori infection. A total of forty patients with non-ulcer dyspepsia and H. pylori infection were randomized to receive either Rabeprazole 10 mg b.i.d. and Amoxicillin 1000 mg t.i.d., for 14 days (R10A), or high-dose Rabeprazole 20 mg twice a day (b.i.d.) and Amoxicillin 1000 mg three times a day (t.i.d) (R20A) for 14 days. H. pylori strains were isolated and antibiotic resistance was measured by the twofold agar dilution method. H. pylori eradication was assessed by 13C-urea breath test at 4 weeks after treatment.

ELIGIBILITY:
Inclusion Criteria:

Patients aged from 18 to 70 years, who presented with upper gastrointestinal symptoms and endoscopically proven H. pylori-positive non-ulcer dyspepsia, were recruited into the study.

Exclusion Criteria:

* patients with peptic ulcer,
* previous H. pylori eradication treatment,
* previous gastric surgery,
* pregnancy,
* lactation,
* major systemic diseases,
* receipt of anti-secretory therapy,
* antibiotics or bismuth in the preceding four weeks, or - allergy to any one of the medications in the regimen.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-04; Primary Completion 2011-10 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
13C-urea breath test | 4 weeks after treatment
  When the outcome of 13C-urea breath test is more than 4%, the helicobacter pylori infection is still exist(positive).

SECONDARY OUTCOMES:
antibiotic resistance | 3 weeks
  H. pylori strains were isolated and antibiotic resistance was measured by the twofold agar dilution method.Minimal inhibitory concentrations (MIC) of Metronidazole (Met), Clarithromycin (Cla), and Amoxicillin (Amo) were determined.MIC of Met>8ug/ml, Cla>2ug/ml, Amo>8ug/ml were determined as resistance breakpoints

CONTACTS AND LOCATIONS:
Overall Officials: Li X B, M.D., Ph.D., Study Chair — Shanghai Jiao-Tong University School of Medicine Renji Hospital
Locations (1):
- GI Division, Shanghai Jiao-Tong University School of Medicine Renji Hospital, Shanghai, Shanghai Municipality, China